CLINICAL TRIAL: NCT07399535
Title: Clinical Investigation of Herbal Formulation and Its Efficacy in Polycystic Ovarian Syndrome
Acronym: PCOS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Saba Zubair, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2024-GENL/101/JPMC; NO.F.2-81/2024-GENL/101/JPMC (Other: Jinnah Postgraduate Medical Centre Karachi)
Record Dates: First submitted 2025-12-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Herbal Medicine; Infertility; Metabolic Disorder
Keywords: polycystic ovarian syndrome; herbal formulation; infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Metabolic Diseases | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Herbal formulation treated group (Experimental): Herbal formulation 500 mg twice daily for 4 months in PCOS patients
  Interventions: Drug: Herbal Formulation
- Metformin XR treated group (Active Comparator): Metformin XR 750 mg twice daily for 4 months in PCOS patients
  Interventions: Drug: Metformin XR
- Adjunct Group (Experimental): Herbal formulation 500 mg and Metformin XR 750 mg twice daily for 4 months in PCOS patient
  Interventions: Drug: Metformin 750 mg and herbal formulation 500 mg

INTERVENTIONS:
Drug: Herbal Formulation — Herbal Formulation 500mg twice daily for 4 months in PCOS patients
  Other Names: Melats P
  Arms: Herbal formulation treated group
Drug: Metformin XR — Metformin XR 750mg twice daily for 4 months in PCOS patients
  Other Names: Glucophage
  Arms: Metformin XR treated group
Drug: Metformin 750 mg and herbal formulation 500 mg — Herbal formulation and Metformin twice daily for 4 months in PCOS patients
  Arms: Adjunct Group

SUMMARY:
Polycystic Ovarian Syndrome (PCO) is a metabolic disorder that afflicts the women of childbearing age. An approximate of 5-10% women are the victim of this disorder. PCOS is a leading cause of infertility in females these days and is characterized by Hyperandrogenism, Chronic Anovulation, Impaired fertility, obesity, Hirsutism, Acne, Obesity, Metabolic disturbances (dyslipidemias, Hyperinsulinemia, insulin resistance, and type- 2 diabetes), and Endometrial Hyperplasia. This study will test a combination of herbal medications (Melats P) in women with PCOS to determine which works best to overcome infertility.

DETAILED DESCRIPTION:
Polycystic Ovarian Syndrome is a point of concern these days in female population around the world.The patients feel psychological and mentally unhealthy. PCO effects around 6- 14% of women worldwide. PCOS is characterized by hormonal dis-regulation and hyperinsulinemia. Improvements in sex hormones and insulin sensitivity in PCOS women, either through lifestyle changes or through pharmaceutical intervention, have consistently resulted in a marked improvement in the reproductive and metabolic abnormalities in PCOS Commonly prescribed treatment for PCOS include oral contraceptives (OCPs), metformin, pioglitazone, estrogen, GnRH agonist, myo-inositol, letrozole and clomiphene citrate. Despite their effectiveness in symptom relief and ovulation induction, these treatments are associated with adverse effects including weight gain, cardiac issues, lactic acidosis, dysmenorrhea, and abdominal discomfort (Hussain et al., 2022). Given the limitations of conventional drugs, Herbal therapies are gaining attention for their multi-targeted ability to restore natural hormonal balance, improve ovulation and offer symptom relief with minimal side effects (Hussain et al., 2022). In this context, the present study is designed to explore the therapeutic benefits of a novel polyherbal formulation that includes Momordica charantia L., Linum usitatissimum, Symplocos racemose bark, Allium cepa L., Tribulus terrestris, and eggshell. These ingredients were selected based on their various pharmacological properties that are relevant to the pathophysiology of PCOS. This study will evaluate the safety and effectiveness of Melats P in achieving a successful menstruation regulation in PCOS women.We will recruit 3 groups , First group with conventional treatment (Metformin ) , Second with Alternative medicine having a herbal Formulation ( Melats P) and Third group patients will receive both Conventional (Metformin) and Herbal Formulationn (Melats P).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of reproductive age (18-40 years).
* Subjects with a diagnosis of polycystic ovary syndrome (PCOS) confirmed by clinician diagnostic criteria.
* Subjects with insulin resistance defined as HOMA-IR > 2.00.

Exclusion Criteria:

* Pregnant or lactating women.
* Subjects with known Cushing's syndrome.
* Subjects with late-onset congenital adrenal hyperplasia.
* Subjects with androgen-secreting tumors.
* Subjects with uncontrolled thyroid disease.
* Subjects with hyperprolactinemia.
* Subjects with diabetes mellitus.
* Subjects with uncontrolled hypertension.
* Subjects with other cardiovascular diseases.
* Subjects with acute or chronic infections.
* Subjects with any known malignancy.
* Subjects with impaired renal function (serum creatinine > 1.5 × ULN).
* Subjects with impaired liver function (serum ALT ≥ 2.5 × ULN).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female subjects in reproductive age (i.e. 18-40 years)
Enrollment: 116 (Estimated)
Dates: Start 2025-02-22 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Regulation of Menstrual Cycle | Baseline to 4 months
  Improvement and restoration of regular ovulatory menstrual cycles ( cycle length 21-35 days) after 4 months of treatment, assessed through menstrual history and ultrasonographic confirmation of ovulation. Ovulation confirmed by transvaginal ultrasonography, defined by the presence of a dominant follicle followed by follicular rupture during the treatment period.

SECONDARY OUTCOMES:
Serum Follicle-Stimulating Hormone (FSH) Levels | Baseline and after 4 months
  Change in serum follicle-stimulating hormone (FSH) concentration measured using standard laboratory assays. Unit of Measure: mIU/mL, Normal Range: Women (Follicular Phase): 3.5 - 12.5 , Women (Ovulation Phase): 4.7 - 21.5, Women (Luteal Phase): 1.7 - 7.7
Serum Luteinizing Hormone (LH) Levels | Baseline and after 4 months
  Change in serum luteinizing hormone (LH) concentration measured using standard laboratory assays. Unit of Measure: mIU/mL, Normal Range: Women (Follicular Phase): 1.9 - 9.2, Women (Ovulation Phase): 6.1 - 49.1, Women (Luteal Phase): 1.3 - 10.8
Serum Testosterone Levels | Baseline and after 4 months
  Change in serum testosterone levels measured using standard laboratory assays. Unit of Measure: ng/mL, Normal Range: 18-49 years: 0.084-0.481
Glycated Hemoglobin (HbA1c) Level | Baseline and after 4 months
  Change in glycated hemoglobin (HbA1c) percentage measured using standardized laboratory methods. Unit of Measure: %, Normal Range: Normal <5.6%, Prediabetes: 5.7% - 6.4%, Diabetes: 6.5% or higher
Fasting Serum Insulin Concentration | Baseline and after 4 months
  Change in fasting serum insulin concentration measured using standard laboratory assays. Unit of Measure: µIU/mL, Normal Range: 2 to 25
HOMA-IR | Before and after 4 months
  HOMA-IR will be calculated before and immediately after 90-day treatment. HOMA-IR is calculated using the following equation: HOMA-IR = fasting plasma glucose in mmol/L×fasting insulin in μU/ml/22.5.
Body Weight | Baseline and after 4 months
  Change in body weight measured using a calibrated weighing scale. Unit of Measure:
  kg

OTHER OUTCOMES:
Assessment of quality of life via Polycystic Ovary Syndrome Quality of Life scale (PCOSQOL) | Before and after 4 months
  The Polycystic Ovary Syndrome Quality of Life Scale (PCOSQOL) is a disease-specific questionnaire used to assess the impact of polycystic ovary syndrome on quality of life. It evaluates five domains: Emotions (8 items), Body Hair (5 items), Weight (5 items), Infertility Problems (4 items), and Menstrual Problems (4 items). Cronbach's alpha were above 0.7 when the PCOSQL was validated (Jones et al., 2004). It has 26 items and uses a 7-point Likert-type scale.
  Scale Range:
  Minimum value: 1 Maximum value: 7
  Lower scores indicate decreased quality of life, while higher scores indicate improved quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Zubair, PhD scholar, Principal Investigator — University of Sindh Jamshoro
Locations (1):
- Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kartal S, Tsintsadze LN, Berezhiani VI VI. Localized structures of electromagnetic waves in hot electron-positron plasmas. Phys Rev E Stat Phys Plasmas Fluids Relat Interdiscip Topics. 1996 Apr;53(4):4225-4228. doi: 10.1103/physreve.53.4225. No abstract available. PMID 9964744
- [Background] Brolin RE. The antiobstruction stitch in stapled Roux-en-Y enteroenterostomy. Am J Surg. 1995 Mar;169(3):355-7. doi: 10.1016/S0002-9610(99)80175-5. PMID 7879843
- [Background] Thompson GR. Plasma exchange for hypercholesterolaemia. Lancet. 1981 Jun 6;1(8232):1246-8. doi: 10.1016/s0140-6736(81)92412-0. No abstract available. PMID 6112576
- [Background] Duck-Chong CG, Henderson-Smart DJ, Gupta JM, Hensley WJ. Measurement of "lamellar body phospholipid" in amniotic fluid as a method for assessing fetal lung maturity. Clin Chem. 1981 Nov;27(11):1851-5. PMID 6895349
- [Background] Penn I. Primary malignancies of the hepato-biliary-pancreatic system in organ allograft recipients. J Hepatobiliary Pancreat Surg. 1998;5(2):157-64. doi: 10.1007/s005340050027. PMID 9745082
- [Background] Iioka Y, Kikuchi K, Tada H, Isogai S, Urayama T. Plasma soluble fibrin monomer complexes in nephrotic syndrome--with reference to hypoalbuminemia. Tohoku J Exp Med. 1984 May;143(1):53-7. doi: 10.1620/tjem.143.53. PMID 6464012
- [Background] Santos E, Kaback HR. Involvement of the proton electrochemical gradient in genetic transformation in Escherichia coli. Biochem Biophys Res Commun. 1981 Apr 30;99(4):1153-60. doi: 10.1016/0006-291x(81)90739-7. No abstract available. PMID 6266413
- [Background] Usher K, Holmes C. Ethical aspects of phenomenological research with mentally ill people. Nurs Ethics. 1997 Jan;4(1):49-56. doi: 10.1177/096973309700400106. PMID 9052181
- [Background] Poole PM. Continuous bladder drainage. Nurs Mirror Midwives J. 1972 Nov 24;135(21):42-3. No abstract available. PMID 4485297
- [Background] Jones GL, Benes K, Clark TL, Denham R, Holder MG, Haynes TJ, Mulgrew NC, Shepherd KE, Wilkinson VH, Singh M, Balen A, Lashen H, Ledger WL. The Polycystic Ovary Syndrome Health-Related Quality of Life Questionnaire (PCOSQ): a validation. Hum Reprod. 2004 Feb;19(2):371-7. doi: 10.1093/humrep/deh048. PMID 14747184
- [Background] Zegers-Hochschild F, Dickens BM, Dughman-Manzur S. Human rights to in vitro fertilization. Int J Gynaecol Obstet. 2013 Oct;123(1):86-9. doi: 10.1016/j.ijgo.2013.07.001. Epub 2013 Aug 6. PMID 23932062
- [Background] Wasilewski T, Lukaszewicz-Zajac M, Wasilewska J, Mroczko B. Biochemistry of infertility. Clin Chim Acta. 2020 Sep;508:185-190. doi: 10.1016/j.cca.2020.05.039. Epub 2020 May 21. PMID 32446954
- [Background] Norman RJ, Dewailly D, Legro RS, Hickey TE. Polycystic ovary syndrome. Lancet. 2007 Aug 25;370(9588):685-97. doi: 10.1016/S0140-6736(07)61345-2. PMID 17720020
- [Background] Murri M, Insenser M, Fernandez-Duran E, San-Millan JL, Luque-Ramirez M, Escobar-Morreale HF. Non-targeted profiling of circulating microRNAs in women with polycystic ovary syndrome (PCOS): effects of obesity and sex hormones. Metabolism. 2018 Sep;86:49-60. doi: 10.1016/j.metabol.2018.01.011. Epub 2018 Feb 2. PMID 29410349
- [Background] Dickerson EH, Cho LW, Maguiness SD, Killick SL, Robinson J, Atkin SL. Insulin resistance and free androgen index correlate with the outcome of controlled ovarian hyperstimulation in non-PCOS women undergoing IVF. Hum Reprod. 2010 Feb;25(2):504-9. doi: 10.1093/humrep/dep393. Epub 2009 Nov 17. PMID 19920068
- [Background] Azziz R, Woods KS, Reyna R, Key TJ, Knochenhauer ES, Yildiz BO. The prevalence and features of the polycystic ovary syndrome in an unselected population. J Clin Endocrinol Metab. 2004 Jun;89(6):2745-9. doi: 10.1210/jc.2003-032046. PMID 15181052
- [Background] Sidra S, Tariq MH, Farrukh MJ, Mohsin M. Evaluation of clinical manifestations, health risks, and quality of life among women with polycystic ovary syndrome. PLoS One. 2019 Oct 11;14(10):e0223329. doi: 10.1371/journal.pone.0223329. eCollection 2019. PMID 31603907
- [Background] Shakil M, Ashraf F, Wajid A. Sexual functioning as predictor of depressive symptoms and life satisfaction in females with Polycystic Ovary Syndrome (PCOS). Pak J Med Sci. 2020 Nov-Dec;36(7):1500-1504. doi: 10.12669/pjms.36.7.2562. PMID 33235564